CLINICAL TRIAL: NCT01859585
Title: Comparing the Efficacy of Parecoxib and Ketorolac as Preemptive Analgesia in Patients Undergoing Posterior Lumbar Spinal Fusion
Brief Title: Efficacy Parecoxib and Ketorolac as Preemptive Analgesia in Spine Fusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, KOOPONG SIRIBUMRUNGWONG, MD, Comparing the efficacy of Parecoxib and Ketorolac as preemptive analgesia in patients undergoing posterior lumbar spinal fusion, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PSU-0001
Record Dates: First submitted 2013-05-15; First posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Postoperative Pain
Keywords: preemptive analgesia; lumbar fusion; Parecoxib; Ketorolac
MeSH Terms: conditions — Pain, Postoperative | interventions — parecoxib; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Parecoxib (Experimental): Parecoxib
  Interventions: Drug: Parecoxib
- Ketorolac (Experimental): Ketorolac
  Interventions: Drug: Ketorolac
- No medication (No Intervention): No medication

INTERVENTIONS:
Drug: Parecoxib — Parecoxib 40 mg intravenous
  Other Names: Dynastat
  Arms: Parecoxib
Drug: Ketorolac — Ketorolac 30 mg intravenous
  Other Names: Ketolac
  Arms: Ketorolac

SUMMARY:
The purpose of this study is to evaluate the efficacy of Parecoxib and Ketorolac as a preemptive analgesia in patients undergoing lumbar spinal fusion.

DETAILED DESCRIPTION:
A prospective, double-blinded randomized control trial. Randomly allocated patient undergoing posterior lumbar spinal fusion into 3 groups (n=32) to receive Parecoxib, Ketorolac and Placebo around 30 minutes prior to incised skin. Efficacy was assessed by visual analog scale score (0-10), total opioid consumption, complication and bleeding also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lumbar spinal fusion for one to three levels
* ASA class I or II

Exclusion Criteria:

* History of allergy to Sulfa group
* History of allergy to OPOID or NSAIDs
* Contraindicate to NSAIDs use
* History of coagulopathy or platelet disfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2011-03; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Pain score | Postoperative time up to 24 hours
  recorded as Verbal Numerical Rating Scare 0-10

SECONDARY OUTCOMES:
Total amount of opioid consumption postoperatively | Postoperative 24 hours

OTHER OUTCOMES:
Amount of drain output and Other Adverse effect | 7 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Koopong Siribumrungwong, MD, Principal Investigator — Orthopedic Department, Faculty of Medicine, Prince of Songkla University, Songkla, Thailand
Locations (1):
- Faculty of Medicine, Prince of Songkla University, Hadyai, Sonkla, Thailand

REFERENCES:
- [Derived] Siribumrungwong K, Cheewakidakarn J, Tangtrakulwanich B, Nimmaanrat S. Comparing parecoxib and ketorolac as preemptive analgesia in patients undergoing posterior lumbar spinal fusion: a prospective randomized double-blinded placebo-controlled trial. BMC Musculoskelet Disord. 2015 Mar 18;16:59. doi: 10.1186/s12891-015-0522-5. PMID 25886746